CLINICAL TRIAL: NCT01716624
Title: A Pilot Study Comparing the Effects of Botulinum Toxin A and Standard Oxybutynin Therapy as First Line Treatment for the Poorly Compliant Pediatric Neurogenic Bladder
Brief Title: Botox Versus Oxybutynin as First Line Treatment for the Poorly Compliant Pediatric Neurogenic Bladder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Sumit Dave, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R-11-140; 17787 (Other: REB)
Record Dates: First submitted 2011-06-29; First posted 2012-10-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Neurogenic Bladder
Keywords: Pediatric
MeSH Terms: conditions — Urinary Bladder, Neurogenic | interventions — oxybutynin; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxybutynin (Active Comparator)
  Interventions: Drug: Oxybutynin
- Botulinum Toxin A injection (Experimental)
  Interventions: Drug: Botulinum Toxin A injection

INTERVENTIONS:
Drug: Oxybutynin — standard oral therapy
  Arms: Oxybutynin
Drug: Botulinum Toxin A injection — 10 units/kg injected into the detrusor muscle using cystoscopy
  Arms: Botulinum Toxin A injection

SUMMARY:
The purpose of this study is to investigate the use of Botulinum Toxin A as primary therapy for children with neurogenic bladder due to spina bifida and compare results with standard oral oxybutynin therapy. This study hopes to demonstrate that Botulinum Toxin A can maintain or improve bladder storage function without side effects associated with oxybutynin use.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spina bifida and neurogenic bladder
* Performing clean intermittent catheterization (CIC)
* Taking 0.3-0.4 mg/kg/day of oxybutynin for a poorly compliant bladder
* Has not had previous bladder surgery
* Has had a urodynamic or videourodynamic study done within the last 6 months
* Upper motor neuron (UMN) type bladder demonstrated on last urodynamic study
* Urodynamic study (UDS) showing either detrusor leak point pressure >40cm H2O; 30cm below capacity <60% of total bladder capacity, 20 cm capacity <70% of bladder capacity
* Able and willing to complete CIC Diaries and Quality of Life Questionnaires
* Consent and assent given to participate in trial

Exclusion Criteria:

* History of lung disease, recurrent aspiration or severe neurological impairment which may increase risk of Botox toxicity or anesthesia
* Positive urine culture
* Known allergy to Botox

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To assess urodynamic effects of intravesical botulinum toxin A injection to standard oral dose therapy | Primary outcomes will be assessed at 3 and 6 months
  The following urodynamic parameters will be measured;
  1. Change in end fill pressure or detrusor leak point pressure (cm H2O)
  2. Change in 20 and 30 cm H2O below volumes expressed as percentage of bladder capacity
  3. Change in reflex volume (percentage of bladder capacity at which neurogenic detrusor overactivity starts)

SECONDARY OUTCOMES:
Calculate accrual rate | Secondary outcomes will be assessed at 6 months
Calculate cross over rate | Secondary outcomes will be assessed at 6 months
Calculate adverse event rates | Secondary outcomes will be assessed at 6 months
Compare the side effects of standard oral therapy compared to Botulinum toxin A injection | Secondary outcomes will be assessed at 6 months
Calculate drop out rate | Secondary outcomes will be assessed at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sumit Dave, MD, Principal Investigator — London Health Sciences Centre, Laweson Health Research Institute
Locations (1):
- London Health Sciences Centre - Victoria Hospital, London, Ontario, Canada